CLINICAL TRIAL: NCT05639049
Title: Capsular Bag Performance of Two Hydrophobic Intraocular Lenses of Different Design
Brief Title: Performance of Two Hydrophobic IOLs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Enova
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Cataract
Keywords: Cataract; Cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enova GF3 (Experimental): Patient will receive the monofocal IOL in one eye during cataract surgery
  Interventions: Device: Enova GF3
- Tecnis 1-piece ZCB00 (Experimental): Patient will receive the monofocal IOL in one eye during cataract surgery
  Interventions: Device: Tecnis 1-piece ZCB00

INTERVENTIONS:
Device: Enova GF3 — Enova GF3, monofocal IOL
  Arms: Enova GF3
Device: Tecnis 1-piece ZCB00 — Tecnis 1-piece ZCB00, monofocal IOL
  Arms: Tecnis 1-piece ZCB00

SUMMARY:
Comparison of the capsular bag performance of two hydrophobic intraocular lenses of different design.

DETAILED DESCRIPTION:
Continuous improvements in cataract surgery technique, intraocular lens (IOL) materials, and design over the past few decades, have led to a more safe procedure with satisfactory refractive outcomes and a short rehabilitation time. By that, patients' expectations concerning their postoperative visual quality and refractive outcome are increasing. However, two main problems might occur after cataract surgery: instability of the IOL position in the capsular bag and formation of posterior capsule opacification (PCO). Both may decrease the optical performance of an IOL.

The performance of an IOL depends on its behaviour in the capsular bag, which has an influence on the anterior chamber depth (ACD), as well as the postoperative refractive shift, the tilt and decentration of the IOL. Several factors such as IOL design and material, capsulorhexis size, capsular bag diameter, and capsular fibrosis or shrinkage may lead to a suboptimal IOL position. Misalignment of an IOL away from the retina leads to a myopic shift, while towards the retina leads to a hyperopic outcome. This explains why inaccurate prediction of postoperative ACD remains the main source of error in IOL power calculation.

One main goal of modern cataract surgery is to yield a low and predictable ACD shift as well as low degrees of IOL tilt and decentration after surgery in order to achieve ideal optical performance of the IOL.

Another aspect of capsular bag performance of an IOL is posterior capsule opacification (PCO). PCO is one of the most frequent long-term complications after cataract surgery leading to dissatisfying results by decreased visual function. Source of PCO are lens epithelial cells from the equator of the lens capsule, which acquire the ability to migrate and proliferate, causing epithelial ingrowth between the IOL and the posterior capsule. It is estimated that PCO occurs at a rate of 12% one year, 21% three years, and 28% five years after cataract surgery. PCO can be treated with neodymium-doped yttrium aluminium garnet (Nd:YAG) laser capsulotomy. However, complications including an increase in intraocular pressure, ocular inflammation, cystoid macular edema, and retinal detachment may occur after this treatment. Hence lower rates of PCO would improve patients long term safety following cataract surgery. Moreover, it would increase patient satisfaction.

The material and design of an IOL may have an effect on the formation of PCO. Sharp optic edge design has been shown to be a major factor in the prevention of PCO. Furthermore, acrylic and silicone hydrophobic materials showed a lower risk for PCO formation and lower rates of postoperative Nd:YAG laser capsulotomy than hydrophilic IOLs.

In this study the ACD shift and IOL tilt and centration as well as the PCO formation of an IOL with a new design, the Enova GF3 IOL will be compared to a standard monofocal IOL, the Tecnis 1-piece ZCB00.

90 eyes of 45 patients will be included into this study. According to the randomization, the ENOVA GF3 will be implanted in one eye and the ZCB00 in the fellow eye of each patient. Follow-up visits will take place 1 week, 3 months, 6 months, and 12 months after the surgery. At each visit a slitlamp examination, non-contact intraocular pressure measurement, refraction, visual acuity testing, biometry, retroillumination photography, and purkinjemeter assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age-related bilateral cataract
* Age 21 or older
* Visual acuity > 0.05
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Written informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome (PEX), traumatic cataract, intraoperative Floppy Iris Syndrome (IFIS), or other co-morbidities that could affect capsular bag stability (e.g. Marfan syndrome)
* Any ophthalmic comorbidity that may compromise visual function or create problems with measurements (e.g. macular degeneration, amblyopia, corneal scars, etc.)
* Previous ocular surgery or trauma
* Pregnancy (pregnancy test will be taken in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Anterior chamber depth | 24 months
  Anterior chamber depth will be assessed using a biometry device and will be compared between both monofocal IOLs

SECONDARY OUTCOMES:
IOL tilt | 24 months
  IOL tilt will be assessed using the purkinjemeter and will be compared between both IOLs
Posterior capsule opacification (PCO) | 24 months
  PCO will be assessed using retroillumination photography and will be compared between both groups
Visual acuity | 24 months
  Visual acuity will be assessed in the far and intermediate distance using ETDRS charts and will be compared between both groups
Catquest 9SF questionnaire | 24 months
  The Catquest 9SF questionnaire will be handed out to all patients

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided